CLINICAL TRIAL: NCT01945450
Title: Prophylactic Antibiotics for Manual Removal of Retained Placenta in Vaginal Birth
Brief Title: Prophylactic Antibiotics for Manual Removal of Retained Placenta in Vaginal Birth: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0186-HMO-CTIL
Record Dates: First submitted 2013-09-15; First posted 2013-09-18 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-08

CONDITIONS: Endometritis
MeSH Terms: conditions — Endometritis | interventions — Antibiotic Prophylaxis; Ampicillin; Gentamicins; Clindamycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antibiotic prophylaxis (Active Comparator): antibiotic prophylaxis as following: 24 hours coverage with Ampicillin 2 grams*4, Gentamycin 240 mg*1, Clindamycin 600 mg*3
  Interventions: Drug: Antibiotic prophylaxis; Drug: Ampicillin; Drug: Gentamycin; Drug: Clindamycin
- No treatment (No Intervention): No antibiotics

INTERVENTIONS:
Drug: Antibiotic prophylaxis — antibiotic prophylaxis as following: 24 hours coverage with Ampicillin 2 grams*4, Gentamycin 240 mg*1, Clindamycin 600 mg*3
  Arms: Antibiotic prophylaxis
Drug: Ampicillin
  Arms: Antibiotic prophylaxis
Drug: Gentamycin
  Arms: Antibiotic prophylaxis
Drug: Clindamycin
  Arms: Antibiotic prophylaxis

SUMMARY:
Background: There is scarce evidence regarding the necessity of antibiotic prophylaxis in manual revision of the uterus after labor in cases of residual placenta.

Methods: a randomized control trial in which parturients for which the placenta was not separated or there is a suspected residual placenta will be divided randomly to two groups: (1) Revision of uterus or Manual lysis without antibiotic prophylaxis; (2) Revision of uterus or Manual lysis with antibiotic prophylaxis as following: 24 hours coverage with Ampicillin 2 grams*4, Gentamycin 240 mg*1, Clindamycin 600 mg*3. In cases of allergy to Penicillin the antibiotic regimen will be: Gentamycin 240 mg*1, Clindamycin 600 mg*3.

Outcomes: Puerperal fever, endometritis, length of hospitalization after labor, recurrent hospitalization in the first 2 weeks after discharge.

ELIGIBILITY:
Inclusion Criteria:

* suspected retained placenta

Exclusion Criteria:

* Intrapartum fever

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Endometritis rate | 3 years

SECONDARY OUTCOMES:
Puerperal fever | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel